CLINICAL TRIAL: NCT04839471
Title: BI-754091 and Afatinib for Refractory Esophageal Squamous Cell Carcinoma (BEAR Study): a Single-arm, Phase II Study
Brief Title: BI-754091 and Afatinib for Refractory Esophageal Squamous Cell Carcinoma (BEAR Study)
Acronym: BEAR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Health Research Institutes, Taiwan (Other)
Collaborators: Taipei Veterans General Hospital, Taiwan (Other Government); Chang Gung Memorial Hospital (Other); China Medical University Hospital (Other); National Cheng-Kung University Hospital (Other); Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T1220; 1200-0320 (Other: Boehringer Ingelheim)
Record Dates: First submitted 2021-03-31; First posted 2021-04-09 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-06

CONDITIONS: Esophageal Squamous Cell Carcinoma (ESCC)
Keywords: immunotherapy; target therapy
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Afatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BI-754091 plus afatinib (Experimental): BI-754091 plus afatinib
  Interventions: Drug: BI-754091 plus afatinib

INTERVENTIONS:
Drug: BI-754091 plus afatinib — Eligible patients will receive BI-754091 240 mg on D1, afatinib 30 mg/day on day 1 to 21 in a 3-week cycle.

SUMMARY:
This is an open-label, single arm, multi-center study, assessing efficacy and safety of BI-754091 in combination with afatinib as treatment in patients with advanced or metastatic ESCC refractory to at least 1 line of systemic treatment (including chemotherapy or radiation therapy).

DETAILED DESCRIPTION:
Esophageal cancer (EsC) is the sixth leading cancer in the world and is a complex disease with heterogenous subgroups. The squamous cell carcinoma subgroup usually involves the upper part of esophagus and typically occurs in mid-age males. Standard treatment for esophageal squamous cell carcinoma (ESCC) utilizes a trimodality approach comprising of surgery (including resection and reconstruction and/or feeding tube support), radiotherapy and chemotherapy. Addition of tyrosine kinase inhibitors has not shown a benefit in advanced or metastatic ESCC. Immunotherapy, especially checkpoint inhibitors that target the PD-1/PD-L1 axis, have demonstrated clinical benefit in phase III trials for head neck squamous cell carcinoma (HNSCC). This led to the anticipation that immunotherapy could also be useful ESCC due to similar histologic cell types, but before the results presented from KEYNOTE-181, no phase III trial have proven such benefit. It must be emphasized that KEYNOTE-180, KEYNOTE-181 and ONO-4538-07 demonstrated efficacy of immune checkpoint inhibitors in ESCC patients were only 14.3-17%; furthermore, USFDA approved pembrolizumab monotherapy for second line treatment in advanced esophageal cancer only with CPS score≧10. Thus, the benefit of immunotherapy in patients with CPS score less than 10 remains uncertain. With effective target therapy and immunotherapy options lacking, there is a huge unmet need for chemotherapy resistant, advanced or metastatic ESCC. In light of a recent retrospective cohort study demonstrating clinical benefit of using pembrolizumab combined with afatinib for refractory HNSCC, the investigators decide to implement the similar regimen (afatinib plus BI704591) in ESCC patients who had failed multiple lines of chemotherapy

ELIGIBILITY:
Inclusion Criteria:

1. histologically confirmed esophagus squamous cell carcinoma (ESCC);
2. metastatic or unresectable disease;
3. previously treated with at least 1 line of platinum based chemotherapy regimens (including cisplatin or carboplatin);
4. Less than 6 months after the most recent treatment, with documented disease progression by imaging studies according to RECIST 1.1 criteria;
5. presence of at least one measurable lesion according to RECIST 1.1. (the measurable lesion cannot be the biopsy lesion)
6. adequate hematopoietic function which is defined as below:

   1. hemoglobin level ≥ 9 g/dL;
   2. absolute neutrophil count (ANC) ≥ 1,500/mm3;
   3. platelet count ≥ 100,000/mm3;
7. adequate hepatic function which is defined as below:

   1. total bilirubin < 2 mg/dL;
   2. Alanine aminotransferase (ALT) ≤ 3 x ULN;
8. adequate renal function: creatinine clearance rate (CCr) ≥ 50 mL/min ((based upon 24-hour urine collection or calculated by Cockroft-Gault formula); < Cockroft-Gault formula > Male: ((140 - age) × weight [kg])/(72 × serum creatinine[mg/dL]) Female: 0.85 x estimate for male
9. age of 20 years or above;
10. ECOG performance status 0-1;
11. life expectancy of at least 12 weeks;
12. ability to take oral medication;
13. ability to understand and willingness to sign a written informed consent document.
14. Subjects with chronic hepatitis B virus infection (HBV surface antigen (HBsAg) positive) must start antiviral therapy with nucleoside analogs (e.g., entecavir or tenofovir, according to current practice guidelines) before start of study drug treatment and maintained throughout the experimental therapy.

Exclusion Criteria:

1. Any investigational treatment, anti-tumour treatment within 4 weeks or within 5 half-life periods (whichever is shorter) prior to the initiation of trial treatment.
2. Major surgery ('major' according to the Investigator's assessment) performed within 12 weeks prior to first trial treatment or planned within 12 weeks after screening, e.g., hip replacement.
3. Any of the following cardiac criteria:

   * Mean resting corrected QT interval (QTc) >470 msec.
   * Any clinically important abnormalities (as assessed by the Investigator) in rhythm, conduction, or morphology of resting ECGs, e.g., complete left bundle branch block, third degree heart block.
   * Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalaemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years-of-age, or any concomitant medication known to prolong the QT interval.
   * Patients with an ejection fraction (EF) <55% or the lower limit of normal of the institutional standard (if the lower limit of normal of institutional standard is higher than 55%) will be excluded. Only in cases where the Investigator (or the treating physician or both) suspects cardiac disease with negative effect on the EF will the EF be measured during screening using an appropriate method according to local standards to confirm eligibility (e.g., echocardiogram, multi-gated acquisition scan). An historic measurement of EF no older than 6 months prior to first administration of trial drug can be accepted provided that there is clinical evidence that the EF value has not worsened since this measurement in the opinion of the Investigator or of the treating physician or both.
4. Known history of human immunodeficiency virus infection.
5. Active autoimmune disease or a documented history of autoimmune disease, except vitiligo or resolved childhood asthma/atopy.
6. Known history of severe hypersensitivity reactions to other mAbs or known hypersensitivity to the trial drugs or their excipients.
7. Known presence of symptomatic central nervous system (CNS) metastases, unless asymptomatic and off corticosteroids and anti-convulsant therapy for at least 2 weeks prior start of treatment.
8. Immunosuppressive corticosteroid doses (>10 mg prednisone daily or equivalent) within 4 weeks prior to the first dose of study treatment.
9. Men who plan to father a child while in the trial and for at least 6 months after the last administration of trial medication.
10. Other malignancy within the past 5 years except for adequately treated basal or squamous cell skin cancer or cervical cancer in situ.
11. Previously treated with any PD-1 inhibitors, PD-L1 inhibitors, or CTLA-4 inhibitors.
12. Previously treated with gefitinib, erlotinib, afatinib, osimertinib.
13. History or known presence of interstitial pneumonia.
14. Presence of grade 2 or above ascites or pleural effusion.
15. Presence of grade 2 or above diarrhea.
16. Presence of mental disease or psychotic manifestation.
17. Active or uncontrolled infection.
18. significant medical conditions that is contraindicated to study medication or render patient at high risk from treatment complications based on investigator's discretion;
19. pregnant women or nursing mothers, or positive pregnancy test for women of childbearing potential. Patients with childbearing potential shall have effective contraception for both the patient and his or her partner during the study.
20. Received a live vaccine within 30 days prior to the first dose of trial treatment. Seasonal flu vaccines that do not contain live virus are permitted.
21. Patients with tracheo-esophageal fistula or broncho-esophagal fistula.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2021-08-06 (Actual); Primary Completion 2023-07-24 (Actual); Study Completion 2024-06-19 (Actual)

PRIMARY OUTCOMES:
ORR (RECIST 1.1) | 2 years
  to evaluate disease objective response rate (ORR) by RECIST 1.1

SECONDARY OUTCOMES:
DoR | 2 years
  to evaluate duration of response
OS | 2 years
  to evaluate overall survival
PFS | 2 years
  to evaluate progression-free survival
ORR (iRECIST) | 2 years
  to evaluate disease objective response rate by iRECIST
DCR | 2 years
  to evaluate disease control rate
To explore the treatment-related adverse events as assessed by CTCAE v5.0 | 2 years
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Tsang-Wu Liu, Study Director — Taiwan Cooperative Oncology Group, NHRI
Locations (4):
- Taiwan (4):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Cheng-Kung University Hospital, Tainan
  - Taipei Veterans General Hospital, Taipei

REFERENCES:
- [Derived] Kao HF, Liao BC, Huang YL, Huang HC, Chen CN, Chen TC, Hong YJ, Chan CY, Chia JS, Hong RL. Afatinib and Pembrolizumab for Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma (ALPHA Study): A Phase II Study with Biomarker Analysis. Clin Cancer Res. 2022 Apr 14;28(8):1560-1571. doi: 10.1158/1078-0432.CCR-21-3025. PMID 35046059